CLINICAL TRIAL: NCT04551677
Title: Collection of Serum Samples From Children 6 Months to < 9 Years of Age Who Received Fluzone® Quadrivalent and Adults ≥ 65 Years of Age Who Received Fluzone® High-Dose Quadrivalent, Influenza Vaccines, 2020-2021 Formulations
Brief Title: Annual Study for Collection of Serum Samples in Children and Older Adults Receiving the 2020-2021 Formulations of Fluzone Quadrivalent Vaccine and Fluzone High-Dose Quadrivalent Vaccine, Respectively
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GRC00101; U1111-1238-1821 (Other: UTN)
Record Dates: First submitted 2020-08-27; First posted 2020-09-16 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Influenza Immunization; Healthy Volunteers
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; Vaccines, Combined

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months (Experimental): Participants aged 6 to <36 months received a 0.5-milliliters (mL) dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 1. Participants for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP), a second dose was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, No Preservative (0.5-mL dose), 2020-2021 formulation
- Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years (Experimental): Participants aged 3 to <9 years received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 1. Participants for whom 2 doses of influenza vaccine were recommended per ACIP, a second dose was administered at Day 28.
  Interventions: Biological: Fluzone Quadrivalent vaccine, No Preservative (0.5-mL dose), 2020-2021 formulation
- Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years (Experimental): Participants aged >=65 years received a 0.7-mL dose of Fluzone High-Dose Quadrivalent vaccine intramuscularly at Day 1.
  Interventions: Biological: Fluzone High-Dose Quadrivalent vaccine (0.7-mL dose), 2020-2021 formulation

INTERVENTIONS:
Biological: Fluzone Quadrivalent vaccine, No Preservative (0.5-mL dose), 2020-2021 formulation — Pharmaceutical form: Suspension for injection in a pre-filled syringe,
  Route of administration: Intramuscular (IM)
  Other Names: Fluzone® Quadrivalent
  Arms: Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months; Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years
Biological: Fluzone High-Dose Quadrivalent vaccine (0.7-mL dose), 2020-2021 formulation — Pharmaceutical form: Suspension for injection in a pre-filled syringe,
  Route of administration: IM
  Other Names: Fluzone High-Dose Quadrivalent
  Arms: Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years

SUMMARY:
Primary Objective:

To provide serum samples (collected from participants before vaccination [Blood Sample 1] and after final vaccination [Blood Sample 2]) to Center for Biologics Evaluation and Research (CBER) for further analysis by the World Health Organization (WHO), Centers for Disease Control and Prevention (CDC), and Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines. In addition, serum samples from adult participants may be further analyzed by the Sponsor to assess breadth of immune response induced by the study vaccines.

DETAILED DESCRIPTION:
Study duration per participant was approximately 28 days for participants 6 months to less than (<) 9 years of age, and 21 days for participants greater than or equal to (>=) 65 years of age, including 1 to 3 visits (1 or 2 vaccination visits) and 1 or 2 telephone calls, depending on study Group.

The aim of study GRC00101 was to obtain serum samples for submission to CBER to aid in the influenza vaccine strain selection process. There were no outcome measures defined in the protocol; however, the number of collected samples was listed as an outcome for disclosure purposes since outcomes were mandatory for study registration.

ELIGIBILITY:
Inclusion criteria :

* Aged 6 months to <9 years or >=65 years of age on the day of first study vaccination (study product administration).
* For participants 6 to <12 months of age, born at full term of pregnancy (>=37 weeks) and with a birth weight >=5.5 pound (lbs) (2.5 kilograms [kg]).
* Informed consent form (ICF) was signed and dated by participants >=65 years of age.
* Assent form was signed and dated by participants 7 to <9 years of age, and ICF was signed and dated by parent(s) or guardian(s) for participants 6 months to < 9years of age.
* Participants and parent/guardian (of participants 6 months to <9 years of age) were able to attend all scheduled visits and to comply with all study procedures.

Exclusion criteria:

- Participation at the time of study enrollment (or in the 30 days preceding the first study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.

Note: Participants were considered eligible for enrollment if no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the participant would complete safety surveillance for the present study.

* Receipt of any vaccine in the 30 days preceding the first study vaccination, or planned receipt of any vaccine before Visit 2 for participants received 1 dose of influenza vaccine or Visit 3 for participants received 2 doses of influenza vaccine.
* Previous vaccination against influenza (in the 2020-2021 influenza season) with either study vaccine or another vaccine.
* Receipt of immune globulins, blood, or blood-derived products in the 3 months preceding planned inclusion.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the 6 months preceding planned inclusion; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the 3 months preceding planned inclusion).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to study vaccine or to a vaccine containing any of the same substances.

Note: The list of vaccine components was included in the Prescribing Information for each study vaccine.

* Thrombocytopenia, which might be a contraindication for IM vaccination, at the discretion of the Investigator.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol abuse or drug addiction.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of planned vaccination or febrile illness (temperature >=100.4 degree [°] Fahrenheit [38.0° Celsius]). A prospective participant not included in the study until the condition had resolved or the febrile event had subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) or in-laws of the Investigator or employee with direct involvement in the proposed study.
* History of serious adverse reaction to any influenza vaccine.
* Personal history of Guillain-Barré syndrome.
* Any condition that in the opinion of the Investigator would pose a health risk to the participant if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of clinically significant developmental delay (at the discretion of the Investigator), neurologic disorder, or seizure disorder.
* Known seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Months to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (2):
- United States (2):
  - Investigational Site Number 8400001, Bardstown, Kentucky
  - Investigational Site Number 8400002, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: GRC00101 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25270&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 16 September 2020 to 10 October 2020 at 2 active sites in the United States.
Pre-assignment Details: A total of 90 participants were enrolled and vaccinated in the study.
Groups:
- Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months: Participants aged 6 to less than (<) 36 months received a 0.5-milliliters (mL) dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 1. Participants for whom 2 doses of influenza vaccine were recommended per Advisory Committee on Immunization Practices (ACIP), a second dose was administered at Day 28.
- Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years: Participants aged greater than or equal to (>=) 65 years received a 0.7-mL dose of Fluzone High-Dose Quadrivalent vaccine intramuscularly at Day 1.
Period: Overall Study
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years | Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years
Started | 29 | 31 | 30
Vaccinated | 29 | 31 | 30
Completed | 29 | 31 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled and vaccinated participants.
Groups:
- Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months: Participants aged 6 to <36 months received a 0.5-mL dose of Fluzone Quadrivalent vaccine, intramuscularly, at Day 1. Participants for whom 2 doses of influenza vaccine were recommended per ACIP, a second dose was administered at Day 28.
- Total: Total of all reporting groups
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years | Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years | Total
Number analyzed (Participants) | 29 | 31 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 31 | 0 | 60
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 30 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 1.65 (0.518) | 5.13 (1.75) | 73.0 (4.03) | 26.6 (33.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 16 | 41
  Male | 16 | 19 | 14 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 0 | 5
  White | 23 | 30 | 30 | 83
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Aged 6 Months to <9 Years Who Provided Serum Samples for Analysis: Groups 1 and 2
Description: Blood samples were collected from participants at first vaccination at Visit 1 (Day 1; pre-vaccination) and at Day 28 after final vaccination either at Visit 2 (Visit 1 + 28 days) for participants who received 1 dose of influenza vaccine; or at Visit 3 (Visit 2 + 28 days) for participants who received 2 doses of influenza vaccine as recommended by ACIP. Collected blood samples were provided to Center for Biologics Evaluation and Research (CBER) for further analysis by World Health Organization (WHO), Centers for Disease Control and Prevention (CDC), and Food and Drug Administration (FDA) to support formulation recommendations for subsequent influenza vaccines.
Time Frame: Visit 1 (Day 1; pre-vaccination) and 28 days post-final vaccination at Visit 2/Visit 3
Population: Analysis was performed on all vaccinated participants i.e. the participants who had received at least 1 dose of the study vaccine. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years
Number analyzed (Participants) | 29 | 31
Participants
  Visit 1 | 29 | 31
  Visit 2: number analyzed (Participants) | 15 | 30
  Visit 2 | 15 | 30
  Visit 3: number analyzed (Participants) | 14 | 1
  Visit 3 | 14 | 1

2. Primary Outcome: Number of Participants Aged >=65 Years Who Provided Serum Samples for Analysis: Group 3
Description: Blood samples were collected from participants at first vaccination at Visit 1 (Day 1; pre-vaccination) and 21 days after vaccination (Visit 2). Collected blood samples were provided to CBER for further analysis by WHO, CDC, and FDA to support formulation recommendations for subsequent influenza vaccines.
Time Frame: Visit 1 (Day 1; pre-vaccination) and 21 days post-vaccination (Visit 2)
Population: Analysis was performed on all vaccinated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years
Number analyzed (Participants) | 30
Participants
  Visit 1 | 30
  Visit 2 | 30

ADVERSE EVENTS:
Time Frame: Serious adverse events data were collected from Visit 1 (Day 1) up to end of the study (i.e., up to Day 21 for adult participants [>=65 years], up to Day 28 for child participants [6 to <9 years] who had received 1 dose and up to Day 56 for participants who had received 2 doses).
Description: Non-serious adverse event data were not planned to be collected in this study. Analysis was performed on all vaccinated participants.
Arm/Group | Group 1: Fluzone Quadrivalent Influenza Vaccine: 6 to <36 Months | Group 2: Fluzone Quadrivalent Influenza Vaccine: 3 to <9 Years | Group 3: Fluzone High-Dose Quadrivalent Influenza Vaccine: >=65 Years
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT04551677/Prot_SAP_000.pdf